CLINICAL TRIAL: NCT05250934
Title: Robotic Telerehabilitation: Feasibility of a Robotic Treatment of the Upper Limb With Remote Supervision in Patients With Stroke
Brief Title: Robotic Telerehabilitation of the Upper Limb in Stroke
Acronym: TELEREHAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Irene Giovanna Aprile, Director of the Neurorehabilitation Department, Neurologist, Principal Investigator, Fondazione Don Carlo Gnocchi Onlus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDG-Telerehab2021
Record Dates: First submitted 2022-02-11; First posted 2022-02-22 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Stroke
Keywords: Robotic rehabilitation; Telerehabilitation; Upper extremity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robotic group (Experimental): In the robotic group, each patient undergoes 20 upper limb robotic telerehabilitation sessions, each session lasting 1 hour. The frequency is 5 sessions/week. Each session is performed at the patient's home, with direct supervision of a caregiver and remote supervision of a physical therapist, using three webcams able to show (a) the frontal and (b) the sagittal plane of the patient, as well as (c) the monitor of the robot.
  Interventions: Device: Robotic rehabilitation

INTERVENTIONS:
Device: Robotic rehabilitation — The upper limb rehabilitation will be carried out with the planar rehabilitation robot Icone (a CE Class IIA medical device manufactured by Heaxel). The proposed exercises require the patient to move a cursor on the screen using the end-effector of the robot to reach specific points (planar reaching exercises). When the patient is able to perform these exercises independently, the robot assists the movement by minimizing the interaction force applied to the hand and limiting itself to acquiring the kinematic and dynamic parameters of the exercise, which are useful in determining the state of motor skills. Icone assist the subject by applying a force to his hand that helps him complete the task in the phases where the patient plans the movement correctly but is unable to complete it. As a result, the system will enable you to perform planar elbow and shoulder movements in active, passive, or active-assisted modes, with visual and acoustic feedback.
  Other Names: Icone (Heaxel)

SUMMARY:
The goal of the study is to investigate the feasibility and the effects of a home-based upper-limb rehabilitation treatment (based on teleconsulting, telemonitoring, and robotic telerehabilitation using the robot Icone and integrated sensors) in patients with stroke.

DETAILED DESCRIPTION:
Stroke is the second leading cause of death, the third leading cause of disability in the world and the leading cause of disability in the elderly. Rehabilitation treatment is a long and costly process, the effectiveness of which is supported by strong scientific evidence. In recent years, technology has spread to the rehabilitation field and, to date, the use of rehabilitation robotics, in addition to conventional treatment, is recommended by some stroke guidelines. The coronavirus pandemic has required a reorganization of rehabilitation services, but also an enhancement of technology as a tool in the rehabilitation field that can allow treatment in compliance with social distancing. Many scientific works have in fact confirmed the usefulness of these approaches to overcome the limits imposed by the pandemic, in particular for the treatment of disabilities in stroke patients.

The rehabilitation robot Icone (CE marked medical device, Class II-A, produced by Heaxel), is a device with certification for home use and therefore suitable for telerehabilitation. The proposed study aims to test the feasibility of rehabilitation treatment in a home setting based on a system of telecounseling, telemonitoring and robotic telerehabilitation using the robot Icone and integrated sensors for patients with stroke, to overcome the limits imposed by the COVID-19 pandemic.

Patients undergo robotic telerehabilitation treatment, carried out at home. The patient is supervised by a caregiver and, remotely, by a multidisciplinary team thanks to the use of webcams and sensors embedded in the robot. The evaluations, through clinical scales and instrumental evaluations, are carried out both in presence (at the enrollment and the end of the study) and remotely (before the first telerobotic rehabilitation session, in the middle and after the last telerobotic rehabilitation session). The study is included in the Regional Smart Specialization Strategy (S3 - Biorobotics for rehabilitation) for business & life continuity and co-financed by the European Union through LazioInnova

ELIGIBILITY:
Inclusion Criteria:

* ischemic or hemorrhagic stroke (verified by MRI or CT);
* time since stroke onset > 3 months
* cognitive abilities adequate to understand the experiments and the follow instructions
* upper limb impairment (Fugl-Meyer Assessment - upper extremity score ≤58);
* presence of a caregiver to supervise the treatment

Exclusion Criteria:

* fixed contractions in the affected limb (ankylosis, Modified Ashworth Scale equal to 4);
* inability to understand the instructions required for the study;
* behavioral disorders that may influence therapeutic activity;
* other orthopedic or neurological diseases
* inability or unwillingness to provide informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2021-08-08 (Actual); Study Completion 2021-08-08 (Actual)

PRIMARY OUTCOMES:
Changes in Fugl-meyer Assessment Upper Extremity motor functioning | Before the intervention, after a 4-week robotic rehabilitation intervention
  It is a stroke-specific, performance-based impairment index. It ranges from 0 (hemiplegia) to 66 points (normal).
Reliability of the remote evaluation of the Fugl-meyer Assessment Upper Extremity motor functioning (FMA) | Before the intervention
  The value of the FMA obtained by means of online observation of the patient will be assessed in terms of reliability with the value obtained by means of direct observation, using the Intraclass Correlation Coefficient.
System Usability Scale | After a 4-week robotic rehabilitation intervention
  It is a self-administered questionnaire to evaluate usability. It ranges from 0 to 100. Higher scores mean better usability.
Technology Acceptance Model (TAM) | After a 4-week robotic rehabilitation intervention
  It is a self-administered questionnaire to evaluate the acceptance of the provided intervention. It comprises several questions rated on a 7-point likert scale.
Likert for Satisfaction | After a 4-week robotic rehabilitation intervention
  Satisfaction will be assessed using a 11-point likert scale. It ranges from 0 to 10. Higher scores mean higher satisfaction.

SECONDARY OUTCOMES:
Changes in Fugl-meyer Assessment Upper Extremity motor functioning | Before the intervention, after a 2-week robotic rehabilitation intervention
  t is a stroke-specific, performance-based impairment index. It ranges from 0 (hemiplegia) to 66 points (normal).
Changes in Fugl-meyer Assessment - Sensory functioning | Before the intervention, after a 2-week robotic rehabilitation intervention
  It is a stroke-specific, sensory impairment index. It ranges from 0 (worse) to 12 points (best).
Changes in Fugl-meyer Assessment - Sensory functioning | Before the intervention, after a 4-week robotic rehabilitation intervention
  It is a stroke-specific, sensory impairment index. It ranges from 0 (worse) to 12 points (best).
Changes in Numeric Rating Scale for pain | Before the intervention, after a 2-week robotic rehabilitation intervention
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale, from 0 (no pain) to 10 (worst pain imaginable).
Changes in Numeric Rating Scale for pain | Before the intervention, after a 4-week robotic rehabilitation intervention
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale, from 0 (no pain) to 10 (worst pain imaginable).
Changes in the Independence Index | Before the intervention, after a 2-week robotic rehabilitation intervention
  It is a kinematic index computed by means of the robotic device. It represent the ratio between the minor and major axes of the ellipse best fitting the hand path in Cartesian coordinates during a circle drawing task.
Changes in the Independence Index | Before the intervention, after a 4-week robotic rehabilitation intervention
  It is a kinematic index computed by means of the robotic device. It represent the ratio between the minor and major axes of the ellipse best fitting the hand path in Cartesian coordinates during a circle drawing task.
Changes in the Area Index [m2] | Before the intervention, after a 2-week robotic rehabilitation intervention
  It is a kinematic index computed by means of the robotic device. It represent the area of the ellipse best fitting the hand path in Cartesian coordinates during a circle drawing task.
Changes in the Area Index [m2] | Before the intervention, after a 4-week robotic rehabilitation intervention
  It is a kinematic index computed by means of the robotic device. It represent the area of the ellipse best fitting the hand path in Cartesian coordinates during a circle drawing task.
Changes in the Path Index [mm] | Before the intervention, after a 2-week robotic rehabilitation intervention
  It is a kinematic index computed by means of the robotic device. It represents the mean distance of the travelled path from the ideal path during a point-to-point (reaching) task
Changes in the Path Index [mm] | Before the intervention, after a 4-week robotic rehabilitation intervention
  It is a kinematic index computed by means of the robotic device. It represents the mean distance of the travelled path from the ideal path during a point-to-point (reaching) task
Changes in the Movement Duration index [t] | Before the intervention, after a 2-week robotic rehabilitation intervention
  It is a kinematic index computed by means of the robotic device. It represents the mean time required to perform a movement during a point-to-point (reaching) task
Changes in the Movement Duration index [t] | Before the intervention, after a 4-week robotic rehabilitation intervention
  It is a kinematic index computed by means of the robotic device. It represents the mean time required to perform a movement during a point-to-point (reaching) task
Changes in the Peak speed index [m/s] | Before the intervention, after a 2-week robotic rehabilitation intervention
  It is a kinematic index computed by means of the robotic device. It represents the maximum value of the speed during a point-to-point (reaching) task
Changes in the Peak speed index [m/s] | Before the intervention, after a 4-week robotic rehabilitation intervention
  It is a kinematic index computed by means of the robotic device. It represents the maximum value of the speed during a point-to-point (reaching) task
Changes in the Mean speed index [m/s] | Before the intervention, after a 2-week robotic rehabilitation intervention
  It is a kinematic index computed by means of the robotic device. It represents the mean value of the speed during a point-to-point (reaching) task
Changes in the Mean speed index [m/s] | Before the intervention, after a 4-week robotic rehabilitation intervention
  It is a kinematic index computed by means of the robotic device. It represents the mean value of the speed during a point-to-point (reaching) task
Changes in the Smoothness index | Before the intervention, after a 2-week robotic rehabilitation intervention
  It is a kinematic index computed by means of the robotic device. It represents the ratio between the mean and the maximum value of the speed during a point-to-point (reaching) task
Changes in the Smoothness index | Before the intervention, after a 4-week robotic rehabilitation intervention
  It is a kinematic index computed by means of the robotic device. It represents the ratio between the mean and the maximum value of the speed during a point-to-point (reaching) task
Changes in the Hold index [m] | Before the intervention, after a 2-week robotic rehabilitation intervention
  It is a kinetic index computed by means of the robotic device. It represents the mean value of the displacement of the end-effector of the robot when the patient is required to hold it in the middle of the workspace against centrifugal forces aimed to move the end-effector toward the targets. It decreases when the patient's strength increases.
Changes in the Hold index [m] | Before the intervention, after a 4-week robotic rehabilitation intervention
  It is a kinetic index computed by means of the robotic device. It represents the mean value of the displacement of the end-effector of the robot when the patient is required to hold it in the middle of the workspace against centrifugal forces aimed to move the end-effector toward the targets. It decreases when the patient's strength increases.
Changes in the Displacement index [m] | Before the intervention, after a 2-week robotic rehabilitation intervention
  It is a kinetic index computed by means of the robotic device. It represents the mean value of the displacement of the end-effector of the robot when the patient is required to move it toward the eight targets against a centripetal force that try to hold it in the middle of the workspace.
  It increases when the patient's strength increases.
Changes in the Displacement index [m] | Before the intervention, after a 4-week robotic rehabilitation intervention
  It is a kinetic index computed by means of the robotic device. It represents the mean value of the displacement of the end-effector of the robot when the patient is required to move it toward the eight targets against a centripetal force that try to hold it in the middle of the workspace.
  It increases when the patient's strength increases.
Reliability of the remote evaluation of the Independence Index | Before the intervention
  The reliability of the index obtained by the patient using the robot at home will be assessed in terms of reliability with the value obtained by the patient using the robot in the clinic, using the Intraclass Correlation Coefficient.
Reliability of the remote evaluation of the Area Index | Before the intervention
  The reliability of the index obtained by the patient using the robot at home will be assessed in terms of reliability with the value obtained by the patient using the robot in the clinic, using the Intraclass Correlation Coefficient.
Reliability of the remote evaluation of the Path Index | Before the intervention, after a 4-week robotic rehabilitation intervention
  The reliability of the index obtained by the patient using the robot at home will be assessed in terms of reliability with the value obtained by the patient using the robot in the clinic, using the Intraclass Correlation Coefficient.
Reliability of the remote evaluation of the Movement Duration index | Before the intervention, after a 4-week robotic rehabilitation intervention
  The reliability of the index obtained by the patient using the robot at home will be assessed in terms of reliability with the value obtained by the patient using the robot in the clinic, using the Intraclass Correlation Coefficient.
Reliability of the remote evaluation of the Smoothness index | Before the intervention
  The reliability of the index obtained by the patient using the robot at home will be assessed in terms of reliability with the value obtained by the patient using the robot in the clinic, using the Intraclass Correlation Coefficient.
Reliability of the remote evaluation of the Peak speed index | Before the intervention
  The reliability of the index obtained by the patient using the robot at home will be assessed in terms of reliability with the value obtained by the patient using the robot in the clinic, using the Intraclass Correlation Coefficient.
Reliability of the remote evaluation of the Mean speed index | Before the intervention
  The reliability of the index obtained by the patient using the robot at home will be assessed in terms of reliability with the value obtained by the patient using the robot in the clinic, using the Intraclass Correlation Coefficient.
Reliability of the remote evaluation of the Hold index | Before the intervention
  The reliability of the index obtained by the patient using the robot at home will be assessed in terms of reliability with the value obtained by the patient using the robot in the clinic, using the Intraclass Correlation Coefficient.
Reliability of the remote evaluation of the Displacement index | Before the intervention
  The reliability of the index obtained by the patient using the robot at home will be assessed in terms of reliability with the value obtained by the patient using the robot in the clinic, using the Intraclass Correlation Coefficient.It increases when the patient's strength increases.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Aprile, D, PhD, Principal Investigator — Fondazione Don Carlo Gnocchi Onlus
Locations (1):
- Fondazione Don Carlo Gnocchi, Santa Maria della Provvidenza Center, Rome, Italy

REFERENCES:
- [Derived] Germanotta M, Mauro MC, Falchini F, Scotto Di Luzio F, Vollero L, Zollo L, Aprile IG. A robotic rehabilitation intervention in a home setting during the Covid-19 outbreak: a feasibility pilot study in patients with stroke. J Neuroeng Rehabil. 2025 Apr 24;22(1):93. doi: 10.1186/s12984-025-01633-9. PMID 40269913